CLINICAL TRIAL: NCT02835300
Title: Mobile Technology and Online Tools to Improve Asthma Control in Adolescents
Acronym: CampAirPilot
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 3-C Institute for Social Development (Industry)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R44HL127826 Pilot; R44HL127826 (NIH)
Record Dates: First submitted 2016-06-27; First posted 2016-07-18 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: Asthma; Adolescents; e-Health; Intervention
MeSH Terms: conditions — Asthma | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CampAir Intervention (Experimental): Adolescents assigned to receive ASMA 2.0 will receive all seven modules over the two month trial, completing one module per week. Adolescents will be assigned one module per week, but will have free access to all completed modules for the duration of the two-month trial. Each module is expected to take between 30-40 minutes to complete, although adolescents will be able to engage with the software for as long as desired.
  Interventions: Behavioral: CampAir
- Information and Referral Control (Active Comparator): Adolescents assigned to the information-and-referral control condition will be provided access to existing generic asthma education websites. They will also be referred to their medical providers for asthma. After the completion of the trial, all participants will receive access to CampAir.
  Interventions: Behavioral: Information and Referral

INTERVENTIONS:
Behavioral: CampAir — CampAir is a dynamic e-learning intervention to help adolescents with uncontrolled asthma to manage their illness and to improve their asthma control. CampAir consists of seven online modules with one module being completed each week over seven weeks. Each module provides a brief introduction to the topics and strategies focused on in that module followed by a set of interactive exercises and games for practice and personalized feedback.
  Arms: CampAir Intervention
Behavioral: Information and Referral — The information and referral comparator condition will provide access to existing generic asthma education websites. They will also be referred to their medical providers for asthma. After the completion of the trial, all participants will have access to CampAir.
  Arms: Information and Referral Control

SUMMARY:
This project will preliminarily validate CampAir, an empirically-based dynamic e-health intervention (based on the evidence-based ASMA) to assist adolescents with uncontrolled asthma to learn how to manage their illness and improve their asthma control. In addition to developing a highly novel product for adolescents with asthma, the research proposed for this project will address unique scientific questions. Despite the high asthma prevalence among adolescents, few interventions have specifically targeted adolescents. This study is innovative in that it is among the few to focus on adolescents, who are often overlooked by the healthcare system. This research will assess factors associated with successful implementation of CampAir, thereby providing new information regarding how e-health interventions can be effectively developed and implemented for use with adolescents with asthma.

DETAILED DESCRIPTION:
Asthma has high prevalence and morbidity among adolescents, especially urban Hispanic and African American teenagers. Despite this, few interventions have specifically targeted adolescents. School-based and web-based asthma interventions have shown to be effective with younger children, yet few have been developed and tested for adolescents. Investigators have developed Camp Air, an engaging dynamic e-learning intervention to help adolescents with uncontrolled asthma to manage their illness and to improve their asthma control. Camp Air consists of seven online modules with one module being completed each week over seven weeks. Each module provides a brief introduction to the topics and strategies focused on in that module followed by a set of interactive exercises and games for practice and personalized feedback. The investigators will conduct a two group randomized pilot trial with up to 80, 9th - 12th graders with uncontrolled asthma in order (a) to assess the preliminary intervention effects of Camp Air, and (b) to evaluate the feasibility and acceptability of Camp Air. In order to evaluate CAMP Air's utility as both a school- and home-based intervention, adolescents will be enrolled from two sites: 1) NYC public schools (n=up to 38), or 2) the national asthma community at large (n=up to 42). Investigators will also evaluate the reach, acceptability, generalizability, and sustainability of Camp Air using the RE-AIM approach. Investigators hypothesize that over one month post-intervention, relative to controls, Camp Air participants will show significantly greater improvement in asthma-related outcomes. Investigators also hypothesize that ratings and software usage indices will demonstrate that Camp Air is a feasible, usable, and acceptable intervention for use with adolescents. Investigators will also explore evidence of a dose-response in which participants who spend more time engaged with the e-training materials show greater positive change.

ELIGIBILITY:
Inclusion Criteria:

* Ages 13 - 18 years
* Prior asthma diagnosis
* Use of a prescribed asthma medication in the past 12 months
* Uncontrolled asthma, defined as (1) daytime symptoms 3+ days per week, (2) night awakenings 1+ nights per week, or (3) 2+ exacerbation events, i.e. 2+ steroid bursts; 2+ emergency department visits, or 1+ hospitalization for asthma.

Exclusion Criteria:

* Co-morbid diseases that affect lung functioning

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Night Wakenings Due to Asthma | To assess change, this measure will be taken: (1) prior to starting the trial (baseline); (2) within two weeks of completing the last module (immediate post-test); and (3) one month after completing their last module (1-month follow-up).
  Adolescent-reported rates of night wakenings due to asthma in the prior 2 weeks.

SECONDARY OUTCOMES:
Urgent Health Utilization | To assess change, this measure will be taken: (1) prior to starting the trial (baseline); (2) within two weeks of completing the last module (immediate post-test); and (3) one month after completing their last module (1-month follow-up)
  Adolescents will report the number of asthma-related emergency department visits, hospitalizations and acute medical visits in the prior 2 months.
Asthma Morbidity | To assess change, this measure will be taken: (1) prior to starting the trial (baseline); (2) within two weeks of completing the last module (immediate post-test); and (3) one month after completing their last module (1-month follow-up)
  Adolescents will report the number of days in the past 2 weeks (1) they experienced symptoms of wheeze, cough, shortness of breath, or chest tightness; (2) they could not carry out normal activities because of asthma; and (3) absences from school due to asthma.
Asthma self-management skills: Attack Management | To assess change, this measure will be taken: (1) prior to starting the trial (baseline); (2) within two weeks of completing the last module (immediate post-test); and (3) one month after completing their last module (1-month follow-up)
  Self-management indices for youth used in prior research will be used to assess attack management
Asthma self-management skills: Symptom Prevention | To assess change, this measure will be taken: (1) prior to starting the trial (baseline); (2) within two weeks of completing the last module (immediate post-test); and (3) one month after completing their last module (1-month follow-up)
  Self-management indices for youth used in prior research will be used to assess symptom prevention.
Asthma self-management skills: Asthma Self-Efficacy | To assess change, this measure will be taken: (1) prior to starting the trial (baseline); (2) within two weeks of completing the last module (immediate post-test); and (3) one month after completing their last module (1-month follow-up)
  Self-management indices for youth used in prior research will be used to assess asthma self-efficacy.
Quality of life (QOL) | To assess change, this measure will be taken: (1) prior to starting the trial (baseline); (2) within two weeks of completing the last module (immediate post-test); and (3) one month after completing their last module (1-month follow-up)
  QOL in the past week will be assessed with the widely used validated Paediatric Asthma Quality of Life Questionnaire (PAQLQ), which has 23 items in 3 domains: (a) symptoms; (b) emotions, including feelings about self and relationships with siblings or friends; and (c) degree of interference with physical activities.
Asthma control | To assess change, this measure will be taken: (1) prior to starting the trial (baseline); (2) within two weeks of completing the last module (immediate post-test); and (3) one month after completing their last module (1-month follow-up)
  Investigators will use Juniper's Asthma Control Questionnaire (ACQ), a 6-item widely used instrument in pediatric research, shown to be sensitive to treatment effects. Respondents rate their symptoms, night awakening and use of bronchodilators over the previous 7 days on a 7-point scale.
Use of medication | To assess change, this measure will be taken: (1) prior to starting the trial (baseline); (2) within two weeks of completing the last module (immediate post-test); and (3) one month after completing their last module (1-month follow-up)
  Adolescents will report the names of their medications, which will be used to determine if oral steroids and controller medications are used; if oral steroids are reported, investigators will also ask how many times they have been used since the last survey to determine the frequency of steroid bursts.
Self-Management subscale of the Asthma Management and Medication Scale (AMMS) | To assess change, this measure will be taken: (1) prior to starting the trial (baseline); (2) within two weeks of completing the last module (immediate post-test); and (3) one month after completing their last module (1-month follow-up)
  Investigators will use the Self-Management subscale of the Asthma Management and Medication Scale (AMMS), a brief, validated self-report instrument that measures asthma adherence behaviors.
Intervention feedback | 2 weeks post intervention
  Adolescents in both conditions will provide feedback regarding their experiences during the trial period. On a 5-point scale (1=Strongly Disagree to 5=Strongly Agree), respondents will rate the degree to which their experience was: (a) useful for increasing knowledge of asthma and asthma-related symptoms; (b) useful for learning self-management skills; (c) helped decrease the impact of asthma on daily activities; (e) valuable for adolescents with asthma; (f) engaging for adolescents; (g) innovative compared to alternatives; (h) better than alternatives. Participants will also be asked to provide written comments, listing specific concerns or problems. Follow-up interviews at school or via telephone by trained research assistants will be conducted to clarify responses and gather additional details, as needed.
Software usage | Weekly for 7 weeks during intervention
  The system will collect usage data throughout the trial to document when and how the website and software are being used. Whenever adolescents access Camp Air, information about that interaction will be captured and time stamped. Usage statistics will be collected via a combination of HTTP access logs and session cookies to document the number of times a given webpage/tool/resource is accessed, amount of time spent in a given activity, and sequence of steps taken to complete a task.
After-Scenario Questionnaire (ASQ) | 2 weeks post intervention
  Adolescents in the intervention condition will evaluate the technology-based product using the After-Scenario Questionnaire (ASQ).
Post-Study System Usability Questionnaire (PSSUQ) | 2 weeks post intervention
  Adolescents in the intervention condition will evaluate the technology-based product using the Post-Study System Usability Questionnaire (PSSUQ).
Technology Acceptance Model (TAM) | 2 weeks post intervention
  Adolescents in the intervention condition will evaluate the technology-based product using the Technology Acceptance Model (TAM) survey.
CampAir Evaluation | 2 weeks post intervention
  Adolescents in the intervention condition will evaluate the technology-based product using a 5-point scale from 1=Not at all to 5=Extremely) the quality of ASMA 2.0 in the following areas: (a) user friendly; (b) easy to navigate; (c) appealing graphic design; (d) easy to follow directions; (e) jargon free; (f) engaging; (g) high quality content; (h) high value content; (i) relevance to real-life; (j) login functions; (k) search functions; and (l) help functions.
Control Condition Material Usage | 2 weeks post intervention
  Adolescents assigned to the information-and-referral control condition will answer six questions to assess their use of the educational resources provided to them during the intervention phase.
Contamination | 2 weeks post intervention
  Adolescents in the control group in the school sample will be asked three questions about their exposure to CAMP Air, while adolescents in the treatment group in the school sample will be asked questions about their discussing the intervention with other teens in the school and/or sharing the materials with them. Adolescents in the community sample will not be asked contamination-related questions.

CONTACTS AND LOCATIONS:
Overall Officials: James Thomas, PhD, Principal Investigator — 3C Institute
Locations (1):
- 3-C Institute for Social Development, dba 3C Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bruzzese JM, George M, Liu J, Evans D, Naar S, DeRosier ME, Thomas JM. The Development and Preliminary Impact of CAMP Air: A Web-based Asthma Intervention to Improve Asthma Among Adolescents. Patient Educ Couns. 2021 Apr;104(4):865-870. doi: 10.1016/j.pec.2020.09.011. Epub 2020 Sep 15. PMID 33004234